CLINICAL TRIAL: NCT02392026
Title: A Multicenter, Open-Label Study to Evaluate the Safety and Tolerability of Metronidazole Vaginal Gel 1.3% in Adolescent Female Subjects With Bacterial Vaginosis
Brief Title: Safety and Tolerability of Metronidazole Gel 1.3%
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Insud Pharma (Industry)
Collaborators: Allergan Sales, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MG1401
Record Dates: First submitted 2015-03-04; First posted 2015-03-18 (Estimated); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Vaginosis, Bacterial
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metronidazole Gel (Experimental): Metronidazole Vaginal Gel
  Interventions: Drug: Metronidazole Gel

INTERVENTIONS:
Drug: Metronidazole Gel — Metronidazole Vaginal Gel 1.3% administered via applicator
  Other Names: Metro Gel

SUMMARY:
Multicenter, open-label study to evaluate safety and tolerability of Metronidazole Vaginal Gel in females 12 to <18 years for the treatment of bacterial vaginosis.

DETAILED DESCRIPTION:
A multicenter, open-label study to evaluate safety and tolerability of Metronidazole Vaginal Gel 1.3% when administered as a single dose in adolescent females (aged 12 to <18 years) for the treatment of bacterial vaginosis.

ELIGIBILITY:
Inclusion Criteria:

* Provide written assent and parent/legal guardian informed consent and authorization to disclose protected health information.
* Post-menarcheal, adolescent female, 12 to <18 years of age at time of Screening/Baseline Visit (Day 1).
* In good general health at Screening visit with no known medical conditions that, in the Investigator's opinion, may interfere with study participation.
* Has negative urine pregnancy test result prior to study treatment initiation.
* Has clinical diagnosis of bacterial vaginosis.
* Agree to abstain from sexual intravaginal intercourse for study duration.
* Willing to avoid alcohol ingestion for 24 hours after administration of test article.
* Agree to refrain from use of intravaginal products for duration of study (e.g. lubricated condoms, tampons, diaphragms, spermicides, feminine deodorant sprays, douches). Intravaginal Uterine Device (IUD) use is acceptable as long as it has been in place for 30 days prior to study enrollment.
* Willing and able to participate in study, make required visits to the study center, and comply with all study requirements including concomitant medication and other treatment restrictions.

Exclusion Criteria:

* Pregnant, lactating, or planning to become pregnant during study period.
* Currently menstruating or anticipate onset of menses during first 9 days of the study.
* Experience a clinically important medical event with 90 days of Screening/Baseline Visit (Day 1).
* Evidence of other infectious causes of vulvovaginal infection or condition that in the Investigator's opinion would confound the interpretation of the study results.
* Severe symptoms of dysuria and/or pruritus, burning or irritation in vulvovaginal area.
* Received systemic or intravaginal antifungal, antibacterial or antiparasitic drugs within 14 days of Screening/Baseline visit (Day 1). Antiviral therapies (non-intravaginal) are acceptable.
* Has taken disulfiram or systemic corticosteroids (oral or injected) within 14 days of Screening/Baseline Visit (Day 1).
* Had sexual intravaginal intercourse within 24 hours of Screening/Baseline (Day 1).
* Demonstrated previous hypersensitivity to metronidazole, either orally or topically administered, or any form of parabens or benzyl alcohol.
* Known primary or secondary immunodeficiency condition/syndrome.
* Being treated or planning to be treated during the study period for cervical intraepithelial neoplasia (CIN) or cervical carcinoma.
* Using anticoagulation therapy with Coumadin (warfarin).
* Previously treated with test article under this protocol.
* Participate in an experimental drug/device trial within the last 30 days before Screening/Baseline Visit (Day 1).
* Is judged by the Investigator to be unsuitable for any reason.

Ages: 12 Years to 17 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2015-08-12 (Actual); Primary Completion 2016-10-05 (Actual); Study Completion 2016-10-05 (Actual)

PRIMARY OUTCOMES:
Number of subjects with treatment-emergent adverse events (AEs), serious AEs, treatment-related AEs and AEs leading to study discontinuation after Metronidazole Vaginal Gel is administered in post-menarcheal, adolescent females with bacterial vaginosis. | up to 10 days
  No serious AEs reported during the completed study
A multicenter open label to evaluate safety and tolerability of metronidazole vaginal gel 1.3% for adolescents female subject with bacterial and vaginosis | up tp 10 days
  Metronidazole Vaginal Gel 1.3% is safe, well tolerated, and efficacious in treating vaginal discharge and odor in adolescent females aged 12 to < 18 years with bacterial vaginosis. The safety and efficacy profiles in this study were consistent with the known safety and efficacy profiles for the adult population and no new safety concerns were identified.

SECONDARY OUTCOMES:
Number of subjects reporting presence of daily vaginal discharge and/or odor following single dose administration of Metronidazole Vaginal Gel 1.3%assessment of the presence of vaginal discharge and odor following single dose administration. | up to 10 days
  no order or smelling observed

CONTACTS AND LOCATIONS:
Overall Officials: Gina Giannantoni-Ibelli, MS, Study Director — Allergan
Locations (8):
- United States (8):
  - Allergan Research Site #318, Long Beach, California
  - Allergan Research Site #324, Paramount, California
  - Allergan Research Site #315, Bardstown, Kentucky
  - Allergan Research Site #314, New Orleans, Louisiana
  - Allergan Research Site #319, Columbus, Ohio
  - Allergan Research Site #322, Dayton, Ohio
  - Allergan Research Site #321, Memphis, Tennessee
  - Allergan Research Site #316, Irving, Texas